CLINICAL TRIAL: NCT04390997
Title: Determination of the Levels of Lipocalin-2 and Semaphorin3A in Gingival Crevicular Fluid in Subjects With Different Periodontal Diseases
Brief Title: Determination of the Levels of Lipocalin-2 and Semaphorin3A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Merve Ceylan, Research Assistant, Izmir Katip Celebi University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2019-TDU-DİSF-0009
Record Dates: First submitted 2020-05-13; First posted 2020-05-18 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Gingivitis; Periodontitis; Periodontal Diseases
Keywords: Periodontal Disease, Non-surgical Periodontal Treatment, GCF
MeSH Terms: conditions — Gingivitis; Periodontitis; Periodontal Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Periodontally Healthy (No Intervention): 20 participants with bleeding on probing less than 10%, probing depths less than 4mm, and no clinical attachment loss which was measured by six sites per tooth
- Gingivitis (No Intervention): 20 participants with bleeding on probing greater than 10%, probing depths less than 4mm, and no clinical attachment loss which was measured by six sites per tooth
- Periodontitis (Other): 20 participants with bleeding on probing greater than or equal to 30%, probing depths greater than or equal to 5mm at least non-adjacent two teeth in each quadrant of the dentition, and clinical attachment loss greater than or equal to 4mm which was measured by six sites per tooth, and radiographic bone loss on the coronal third of root or severe (vertical/ horizontal) bone loss.
  Interventions: Procedure: Non-surgical Periodontal Treatment

INTERVENTIONS:
Procedure: Non-surgical Periodontal Treatment — Non-surgical periodontal treatment includes scaling and root planning by using curettes and ultrasonic devices only in the periodontitis group.
  Arms: Periodontitis

SUMMARY:
The aim of this clinical trial is to investigate the concentrations of Lipocalin-2 and Semaphorin 3A levels in gingival crevicular fluid in subjects with different periodontal diseases. At the same time for the periodontitis group; the purpose of this study is to analyze the correlation of these proteins with clinical parameters at the first and third months after the nonsurgical periodontal treatment.

DETAILED DESCRIPTION:
In our study, gingival crevicular fluid samples will be taken along with the measurement of all oral clinical parameters from sixty systemically healthy volunteers (20 periodontally healthy, 20 gingivitis, and 20 periodontitis). Gingival crevicular fluid samples will be taken again after the nonsurgical periodontal treatment for the periodontitis group in the first and third months. Lipocalin-2 and Semaphorin 3A levels will be determined by an enzyme-linked immunosorbent assay test (ELISA). Subsequent statistical analyses will be used to interpret protein levels among different groups and peridontitis group after the nonsurgical periodontal treatment.

Possible significant differences may illuminate the future work with Lipocalin-2 and Semaphorin 3A. Also, these glycoproteins may help to develop different diagnostic methods or treatment strategies for future periodontal treatments.

ELIGIBILITY:
Inclusion Criteria:

* Being systemically healthy
* Having at least 20 teeth in the dentition, excluding third molars
* Not using alcohol nor smoking
* Not using medications
* Not taking any antibiotics, anti-inflammatory, nor systemic corticosteroid drugs in the last six months
* Not being in the lactation period nor pregnancy

Exclusion Criteria:

* Having any oral or systemic diseases
* Using alcohol or smoking
* Using medications
* Taking any antibiotics, anti-inflammatory, or systemic corticosteroid drugs in the last six months
* Being in the lactation period or pregnancy
* Being treated with periodontal treatment in the last six months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
The level of Lipocalin-2 | 18 months
  Investigating the concentrations of Lipocalin-2 level in gingival crevicular fluid in subjects with different periodontal diseases.
The level of Semaphorin 3A | 18 months
  Investigating the concentrations of Semaphorin 3A leves in gingival crevicular fluid in subjects with different periodontal diseases.

SECONDARY OUTCOMES:
Effects of non-surgical periodontal treatment on the levels of Lipocalin-2 and Semaphorin3A | 18 months
  Analyzing the correlation of Lipocalin-2 and Semaphorin3A with clinical parameters at the first and third months after the nonsurgical periodontal treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Katip Celebi University, Faculty of Dentistry, Izmir, Cigli, Turkey (Türkiye)